CLINICAL TRIAL: NCT03798327
Title: Video-Assisted Palliative Care Intervention for Patients With Advanced Dementia at Home
Brief Title: Palliative Care at Home for Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nathan Goldstein, Professor, Geriatrics and Palliative Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 17-02787; R56AG067045-01 (NIH)
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Dementia
Keywords: Palliative Care; Home-Based Care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Patient - caregiver pairs
Who Masked: Outcomes Assessor
Masking Description: Single blind control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Palliative Care (Experimental): Randomized to Intervention Arm
  Interventions: Behavioral: Home Palliative Care
- Control Arm (No Intervention): Usual Care - Patients will be cared for by the physician who treats their dementia and other illnesses.

INTERVENTIONS:
Behavioral: Home Palliative Care — Patients/caregivers will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
  Arms: Home Palliative Care

SUMMARY:
The proposed project is a randomized controlled trial of a new home-based palliative care program for adults with advanced dementia and their caregivers within the Mount Sinai Health System. Potential subjects will be identified from Mount Sinai records or referred by a Mount Sinai healthcare provider. Patients will only be approached after authorization by their Mount Sinai physician. Participants who consent to enrollment will be randomized to receive the intervention (home-based palliative care program) or usual care (with their nominated Mount Sinai physician). Patients will be enrolled in the study for 6 months.

Effectiveness of the intervention will be determined through assessment of patient and caregiver reported outcomes and abstraction of data from medical records and administrative claims. Impact on the following parameters will be measured: (i) Patient symptoms, quality of life, satisfaction with care, documentation of advanced directives, receipt of care consistent with preferences (ii) Caregiver burden, satisfaction with care, and depression (iii) Healthcare utilization and costs of care.

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to study the impact of a new home based palliative care program on patients' symptoms, quality of life, satisfaction with care, completion of advance care planning documentation and receipt of care consistent with preferences. In addition, the study will examine the impact of this model of care on patient healthcare utilization, including hospitalization, emergency department utilization, and hospice use prior to death. The trial will also include patients' caregivers, in order to examine the impact of the intervention on caregiver burden and prevalence of depression.

Patients randomized to the intervention will be scheduled for an intake visit. This visit will be undertaken by the team's registered nurse and/or social worker, together with a community health worker, and other team members (advanced practice nurse, MD), depending on patients' needs. Visits will combine a combination of video-teleconferencing technology and in person visits. Following this visit, and in conjunction with the nurse practitioner and/or MD, a care plan will be developed to address areas of clinical need highlighted during the intake visit.

Patients in the intervention arm will receive ongoing monitoring and input (telephone-based, video-based, and in-person) from members of the clinical team, dependent on their identified needs. Patients' cases will be discussed at the weekly IDT meeting, as appropriate to the level of clinical need. Patients and caregivers will be provided with access to a 24 hour telephone line, staffed by a Mount Sinai based physician, which acts as an advice line out of hours. These physicians will be able to provide advice to patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Presence of advanced dementia
* Subject has a Mount Sinai physician who authorizes their participation in the study and receipt of the program
* Subject is resident in Manhattan outside of a long term care facility and is not receiving hospice 5.
* Subject has evidence of capacity to benefit from enrollment in palliative care program
* Subject is conversant in English or Spanish
* Subject has capacity to consent or has a caregiver who can provide consent for the patient

Exclusion Criteria:

* Subject has no usual physician within Mount Sinai
* Subject's usual physician doesn't provide authorization to patient participation
* Subject resident outside of Manhattan or in long term care facility or receiving hospice
* Subject is not conversant in English or Spanish
* Subject cannot provide consent or has no caregiver who can provide consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Goldstein, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai St. Luke's, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Estrada LV, Gelfman L, Zhang M, Espino C, Goldstein N. Challenges and solutions of conducting dementia clinical trials: A palliative care at home pilot for persons with dementia. J Am Geriatr Soc. 2024 Aug;72(8):2544-2551. doi: 10.1111/jgs.18966. Epub 2024 May 22. PMID 38777615

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Palliative Care - Patients: Home Palliative Care: Patients will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
- Usual Care - Control Arm - Patients: Usual Care - Patients will be cared for by the physician who treats their dementia and other illnesses.
- Home Palliative Care - Caregiver: Caregivers of patients cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
- Usual Care - Caregiver: Usual Care - Caregivers of patients will be cared for by the physician who treats their dementia and other illnesses.
Period: Overall Study
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients | Home Palliative Care - Caregiver | Usual Care - Caregiver
Started | 14 | 16 | 14 | 16
Completed | 14 | 16 | 14 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Home Palliative Care - Patients: Home Palliative Care: Patients/caregivers will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
- Home Palliative Care - Caregivers: Caregivers of patients cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.
- Usual Care - Caregivers: Usual Care - Caregivers of patients will be cared for by the physician who treats their dementia and other illnesses.
- Total: Total of all reporting groups
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients | Home Palliative Care - Caregivers | Usual Care - Caregivers | Total
Number analyzed (Participants) | 14 | 16 | 14 | 16 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per the planned analyses, totals were calculated separately for participants in the caregiver and patient groups
  years
    Patients: number analyzed (Participants) | 14 | 16 | 0 | 0 | 30
    Patients | 81.9 (0.75) | 83.4 (0.75) |  |  | 82.7 (1.1)
    Caregivers: number analyzed (Participants) | 0 | 0 | 14 | 16 | 30
    Caregivers |  |  | 59.2 (0.85) | 58.0 (0.85) | 58.6 (14.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10 | 12 | 11 | 11 | 44
  Male | 4 | 4 | 1 | 3 | 12
  Missing | 0 | 0 | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 4 | 13
  Not Hispanic or Latino | 7 | 10 | 8 | 9 | 34
  Unknown or Not Reported | 5 | 1 | 4 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 2 | 7
  White | 9 | 9 | 6 | 6 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 6 | 8 | 19
Number of Participants who lives alone [Count of Participants; unit: Participants] | 2 | 4 | 0 | 1 | 7
Highest Education obtained [Count of Participants; unit: Participants]
  Less than high school diploma/GED | 2 | 4 | 0 | 0 | 6
  High school diploma/GED or greater | 6 | 8 | 5 | 6 | 25
  Missing | 6 | 4 | 9 | 10 | 29
Marital Status [Count of Participants; unit: Participants] — Population: Data collected for caregivers only.
  Participants
    number analyzed (Participants) | 0 | 0 | 14 | 16 | 30
    Married |  |  | 6 | 7 | 13
    Divorced |  |  | 1 | 1 | 2
    Single |  |  | 1 | 3 | 4
    Missing |  |  | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Completed the Symptom Management at the End of Life for Dementia Scale (SM-EOLD)
Description: Number of Patients who completed the SM-EOLD Assessment
  Scale: Symptom Management at the End of Life for Dementia - Likert scale, 9 items, each 0-5, (45 total possible score) higher is worse symptoms
Time Frame: Baseline, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients
Number analyzed (Participants) | 14 | 16
Participants
  Baseline Admission | 14 | 16
  3 months | 6 | 5
  6 months | 2 | 7

2. Secondary Outcome: Number of Patients Who Completed the McGill Quality of Life Assessment
Description: Number of Patients who completed the McGill Quality of Life Assessment
  McGill Quality of Life instrument is assessment in the domains of physical symptoms, emotional well-being, social interactions, and an overall global rating.
  Alzheimer's Disease Scale: Quality of Life - Likert scale, 13 items, each 1-4. Total scale from 13- 52. Higher values are more positive scores.
Time Frame: Baseline, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients
Number analyzed (Participants) | 14 | 16
Participants
  Baseline - Admission | 14 | 15
  3 months | 6 | 5
  6 months | 2 | 7

3. Secondary Outcome: Number of Complete of Advance Directives
Description: The Study Team will examine the patient's chart for completion of advanced directives
  Scale: Study Team will examine the patient's chart for completion of advanced directives (yes/no).
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Preference Consistent Care
Description: The Study Team will examine if the care patients receive is concordant with the care they wanted to receive.
  Scale: Simple chart review of whether care received matches stated preferences (yes/no)
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Number of Caregivers Who Completed the Caregiver Zaria Burden Inventory
Description: Number of Caregivers who completed the Caregiver Zaria Burden Inventory
  Zarit Burden Inventory to determine caregiver burden by using a validated structured 22-item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. Each item is on a 5-point scale range from 0 (never) to 4 (always)
  Scale: Zarit Burden Inventory - Likert scale 0-4,total score = 0-88, higher score is more burden
Time Frame: Baseline, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Home Palliative Care - Caregivers | Usual Care - Caregivers
Number analyzed (Participants) | 14 | 16
Participants
  Baseline - admissions | 13 | 13
  3 months | 6 | 3
  6 months | 2 | 5

6. Secondary Outcome: Number of Caregivers Who Completed the FAMCARE-10 Assessment
Description: Number of Caregivers who completed the FAMCARE-10 Assessment
  FAMCARE-10 to assess caregiver satisfaction by using a validated 10-item structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator.
  Scale: FamCare; Likert scale, 0-3, higher is higher satisfaction
Time Frame: Baseline, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Home Palliative Care - Caregivers | Usual Care - Caregivers
Number analyzed (Participants) | 14 | 16
Participants
  Baseline - Admissions | 13 | 13
  3 months | 6 | 3
  6 months | 2 | 5

7. Secondary Outcome: Number of Caregivers Who Completed the Patient Health Questionnaire (PHQ-9)
Description: Number of Caregivers who completed the Patient Health Questionnaire (PHQ-9)
  PHQ-9 to assess Caregiver Depression by using a validated structured 9 item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
  Scale: Patient Health Questionnaire - 9; Likert scale, 0-3, total possible = 0-27; higher is worse depression [Time Frame: 6 months]
Time Frame: Baseline, 3 months, 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Home Palliative Care - Caregivers | Usual Care - Caregivers
Number analyzed (Participants) | 14 | 16
Participants
  Baseline - Admissions | 13 | 14
  3 months | 6 | 3
  6 months | 2 | 5

8. Secondary Outcome: Mean Change in Number of Hospital Admissions
Description: Healthcare Utilization measured from the data warehouse as well as using the Resource Use Instrument (RUI) collected through interviews with patients. assessed by hospital admissions
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: admissions
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients
Number analyzed (Participants) | 14 | 16
admissions | 0 (0.6) | 0.5 (0.7)

9. Secondary Outcome: Hospital Length of Stay
Description: Patient healthcare utilization as assessed by hospital length of stay over the past 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients
Number analyzed (Participants) | 14 | 16
days | 0 (1.7) | 1.3 (2.9)

ADVERSE EVENTS:
Time Frame: Not collected
Description: Not collected
Arm/Group | Home Palliative Care - Patients | Usual Care - Control Arm - Patients | Home Palliative Care - Caregivers | Usual Care - Caregivers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03798327/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03798327/SAP_001.pdf
  • Informed Consent Form (2022-03-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03798327/ICF_002.pdf